CLINICAL TRIAL: NCT05528913
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2, 12-Week Treatment Study With a 10-Week Follow-up Period to Assess the Efficacy and Safety of Benralizumab (Anti-IL5Rα) in Adult Patients With Chronic Prurigo
Brief Title: Benralizumab in Chronic Prurigo - Investigating Clinical Efficacy (BICPIC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Financing has been withdrawn
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Martin Metz, Prof., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEALSZ-2021-001
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Chronic Prurigo
Keywords: Benralizumab in Chronic Prurigo
MeSH Terms: interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: 2:1 (Benralizumab : Placebo)
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Fasenra 60mg s.c. administration
  Interventions: Drug: Fasenra Prefilled Syringe
- Placebo (Placebo Comparator): Placebo s.c. administration
  Interventions: Other: Matching Placebo Solution

INTERVENTIONS:
Drug: Fasenra Prefilled Syringe — Fasenra 60mg s.c. administration at weeks 0,4 and 8
  Other Names: Benralizumab
  Arms: Benralizumab
Other: Matching Placebo Solution — Placebo s.c. administration at weeks 0,4 and 8
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, Phase 2, 12-Week treatment study with a 10-Week Follow-up period to assess the efficacy and safety of Benralizumab (anti-IL5Rα) in adult patients with chronic prurigo (BICPIC)

DETAILED DESCRIPTION:
Chronic Prurigo (CPG) is a skin disease of unknown incidence and prevalence that can occur in all age groups including children, but which is most prevalent in elderly people. CPG was defined as a distinct disease in 2018 by the Task Force Pruritus of the EADV and diagnosis is based on the presence of chronic pruritus, multiple localized or generalized, pruriginous lesions, and the history and/or signs of a prolonged scratching behavior. While CPG is a disease in its own right, the initial causes of chronic pruritus can be manifold and may be of dermatological, systemic, neurological, psychiatric/psychosomatic, multifactorial or of unknown origin. The pruriginous lesions can be skin-colored, pink or red, hyperkeratotic or excoriated, scaling and/or crusted papules and/or nodules and/or plaques. Depending on the predominant clinical phenotype, CPG subtypes have been defined as papular type, nodular type (also called prurigo nodularis), plaque type, umbilicated type or linear prurigo. Of these, the nodular type is the most frequent one. Although CPG patients are sometimes covered in excoriated intensely pruritic nodules, these skin lesions are always secondary to an intense itch-scratch cycle. Thus, an effective treatment of itch will also lead to the disappearance of the skin lesions. The vast majority of CPG patients are resistant to common therapy and desperate for novel treatment options. Consequently, those affected by intensely itchy CPG are dramatically impaired in their quality of life. Currently, there are no approved therapies for the treatment of CPG available.

The study aims to assess the exploratory efficacy and safety of benralizumab, a monoclonal antibody against IL5Rα in adult patients with chronic prurigo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is informed about study procedures and medications and has given written informed consent before any assessment.
2. Patient is able to communicate with the investigator, understands and complies with the requirements of the study.
3. Clinical diagnosis of CPG for at least 6 months with:

   * Severe pruritus with WI-NRS rating ≥ 6 (Mean of the worst daily intensity over the previous 3 days at Screening and over the previous week at baseline [minimum of at least 5 days during the week preceding the baseline visit]).
   * Pruriginous nodular, papular, plaque and/or umbilicated lesions on upper limbs, trunk, and/or lower limbs
   * At least 20 CPG lesions on the entire body with a bilateral distribution
4. Willing and able to complete a daily symptom Diary for the duration of the study and adhere to the study visit schedules.
5. Women of childbearing potential (WOCBP) must agree to use a highly effective method of birth control
6. Negative COVID-19 test

Exclusion Criteria:

1. Chronic pruritus resulting from another active condition other than CPG
2. Unilateral lesions of prurigo (eg, only one arm affected)
3. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
4. Patients who previously received benralizumab
5. Patients with hypersensitivity to any of the excipients of the IMP or history of anaphylaxis to any biologic therapy or vaccine.
6. Any disorder that is not stable in the opinion of the Investigator and could: (a) Affect the safety of the participant throughout the study, (b) Influence the findings of the studies or their interpretations, (c) Impede the participant's ability to complete the entire duration of study.
7. Inability to comply with study and follow-up procedures.
8. Current malignancy, or history of malignancy within the last 5 years
9. Current active liver disease
10. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test
11. Subjects who live in detention on court order or on regulatory action as per local and national law (see §40 subsection 1 sentence 3 no. 4 Arzneimittelgesetz)
12. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
13. Patients with active COVID-19 infection. Patients with symptoms consistent with COVID-19 infection should be tested prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale of the worst itch (WI-NRS) | Week 0 to week 12
  Percent change from baseline in numerical rating scale of the worst itch

SECONDARY OUTCOMES:
Effects on responder rates | 12 weeks
  Effects on responder rates at week 4, 8 and 12 (defined by > 3 point change on WI-NRS)
Pruritus WI-NRS | 12 weeks
  Absolute and Percent change from baseline in weekly average of the maximum pruritus and average pruritus WI-NRS at every week
Prurigo Activity Score (PAS) | 12 weeks
  Change in prurigo activity score (PAS) from baseline to week 4, 8 and 12
Prurigo Control Test (PCT) | 12 weeks
  Change in the overall disease control, as assessed by the prurigo control test (PCT) from baseline to week 4, 8 and 12
Investigator Global Assessment (IGA) | 12 weeks
  Change in Investigator Global Assessment (IGA)-activity from baseline to week 4, 8 and 12
Investigator Global Assessment (IGA)-stage | 12 weeks
  Change in IGA-stage from baseline to week 4, 8 and 12
Change in the patient's quality of life | 12 weeks
  patient's quality of life assessed by ItchyQoL and Dermatology Life Quality index (DLQI)
Numerical rating scale (NRS) of sleep disturbance | 12 weeks
  Effects on sleep disturbance NRS

CONTACTS AND LOCATIONS:
Overall Officials: Martin Metz, Prof., Principal Investigator — Charité University, Berlin, Germany
Locations (3):
- Germany (3):
  - Hautklinik Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Klinik für Dermatologie, Venerologie und Allergologie, Kiel, Schleswig-Holstein
  - Charite University Medicine, Berlin

IPD SHARING:
Plan to Share IPD: No